CLINICAL TRIAL: NCT06416865
Title: A Randomized, Double-blind, Multi-center, Phase III Trial to Evaluate the Efficacy and Safety of AJU-C52 in Compared With C52R1M for Essential Hypertension Patients in Inappropriately Controlled on C52R1L Treatment
Brief Title: Efficacy and Safety of AJU-C52 in Essential Hypertension Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AJU Pharm Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21HT30601
Record Dates: First submitted 2024-05-12; First posted 2024-05-16 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AJU-C52L, AJU-C52 (Experimental): Treatment Period 1: AJU-C52L+C52R1L placebo
  Treatment Period 2: AJU-C52+C52R1M placebo
  Interventions: Drug: AJU-C52L, AJU-C52
- C52R1L, C52R1M (Experimental): Treatment Period 1: C52R1L+AJU-C52L placebo
  Treatment Period 2: C52R1M+AJU-C52 placebo
  Interventions: Drug: C52R1L, C52R1M

INTERVENTIONS:
Drug: AJU-C52L, AJU-C52 — AJU-C52L+C52R1L placebo: Subjects take the investigational products once a day for 2 weeks.
  AJU-C52+C52R1M placebo: Subjects take the investigational products once a day for 6 weeks.
  Arms: AJU-C52L, AJU-C52
Drug: C52R1L, C52R1M — C52R1L+AJU-C52L placebo: Subjects take the investigational products once a day for 2 weeks.
  C52R1M+AJU-C52 placebo: Subjects take the investigational products once a day for 6 weeks.
  Arms: C52R1L, C52R1M

SUMMARY:
A Randomized, Double-blind, Multi-center, Phase III study to evaluate the efficacy and safety of the AJU-C52 compared with the combination of C52R1M in patients with essential Hypertension Patients who have inappropriately controlled on C52R1L treament

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≤19 years.
* Those who voluntarily signed the informed consent to participate in this study.
* A patient diagnosed with essential hypertension or Patients taking hypertension medication
* Those who are eligible for adequate blood pressure criteria during screening tests: Naïve patient-160 mmHg≤MSSBP<200 mmHg and MSDBP<110 mmHg/Patients taking hypertension medication-140 mmHg≤MSSBP<200 mmHg and MSDBP<110 mmHg

Exclusion Criteria:

* At the screening visit (Visit 1), patients had 3 blood pressure measurements in the arm with the higher average MSSBP, those whose maximum and minimum blood pressure differences are MSSBP 20 mmHg and MSDBP 10 mmHg
* Secondary hypertension patients or those with a history of suspected secondary hypertension
* Cardiovascular/cerebrovascular disease
* Those with a history of malignant tumor within 5 years

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2022-06-27 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Changes in MSSBP(mean sitting systolic blood pressure) | 8th week
  Changes in MSSBP(mean sitting systolic blood pressure) at the 8th week afeter administration of investigational products from the baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- AJU Pharm Co., Ltd., Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No